CLINICAL TRIAL: NCT02269033
Title: Redes en Acción: National Patient Navigator Intervention Study
Brief Title: Redes II National Patient Navigator Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Brooklyn Hospital Center (Other); University of Miami Sylvester Comprehensive Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); University of California, San Francisco (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20080535H; U01CA114657 (NIH)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Patient Navigation; Health Disparities; Latinas; Breast Imaging Reporting and Data System, BI-RADS; underserved
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Navigated Latinas (Experimental): Patient navigators provided culturally sensitive support and guidance to Latina women who presented radiologic abnormalities categorized as BI-RADS 3, 4 and 5. Patient Navigators also collected clinical information from the patients' medical charts.
  Interventions: Behavioral: Patient Navigated Latinas
- Non Navigated Latinas (Active Comparator): A convenience sampling approach was used to recruit non navigated Latinas. Eligibility criteria targeted self-identified Latinas at community-based health clinics, aged > 18 years with an abnormal breast screening mammogram resulting in BI-RADS 3, 4 or 5. Controls were chosen by determining eligibility consecutively backwards from the study start date.
  Interventions: Behavioral: Non Navigated Latinas

INTERVENTIONS:
Behavioral: Patient Navigated Latinas — Patient navigators provided culturally sensitive support and guidance to Latina women who presented radiologic abnormalities categorized as BI-RADS 3, 4 and 5. Patient Navigators also collected clinical information from the patients' medical charts.
  Arms: Patient Navigated Latinas
Behavioral: Non Navigated Latinas — A convenience sampling approach was used to recruit non navigated Latinas. Eligibility criteria targeted self-identified Latinas at community-based health clinics, aged > 18 years with an abnormal breast screening mammogram resulting in BI-RADS 3, 4 or 5. Controls were chosen by determining eligibility consecutively backwards from the study start date.
  Arms: Non Navigated Latinas

SUMMARY:
The purpose of this study is to assess the efficacy of a "patient navigator" program that uses a trained community lay health worker to assist Hispanic patients in utilizing cancer care services. This study is a two part study. The first part of the study consists of a retrospective data collection procedure called "baseline clinical chart audit" of 50 Hispanic women over 18 years of age who have had a mammography abnormality classified as BI-RADS 3, 4 or 5. These data will be drawn from the study clinic's existing records and will serve as baseline data for subjects recruited during the course of the study. The second part of the study, the intervention group, involves the recruitment of 50 low-income, Hispanic women who receive abnormal breast cancer screening results (also classified as BI-RADS 3, 4 or 5) from screening services at local community health clinics. Participants will have significantly higher compliance rates and significantly shorter time lags and between an abnormal screening result, and confirmatory screening tests and commencement of treatment, compared to our baseline. The investigators expect at least a 12% increase in after-screening compliance rate and a 25% reduction in time lags in the treatment group, in relation to the pre-intervention baseline assessment.

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer-related deaths in Latinas, chiefly because of later diagnosis. The time from screening to diagnosis is critical to optimizing cancer care, yet the efficacy of navigation in reducing it is insufficiently documented. Here the investigators evaluate a culturally sensitive patient navigation program to reduce the time to diagnosis and increase the proportions of women diagnosed within 30 days and 60 days. METHODS. The investigators analyzed 425 Latinas who had Breast Imaging Reporting and Data System (BI-RADS) radiologic abnormalities categorized as BI-RADS-3, BI-RADS-4, or BI-RADS-5 from July 2008 to January 2011. There were 217 women in the navigated group and 208 women in the control group. Women were navigated by locally trained navigators or were not navigated (data for this group were abstracted from charts). The Kaplan-Meier method, Cox proportional hazards regression, and logistic regression were used to determine differences between groups. RESULTS. The time to diagnosis was shorter in the navigated group (mean, 32.5 days vs 44.6 days in the control group; hazard ratio, 1.32; P ¼ .007). Stratified analysis revealed that navigation significantly shortened the time to diagnosis among women who had BI-RADS-3 radiologic abnormalities (mean, 21.3 days vs 63.0 days; hazard ratio, 2.42; P < .001) but not among those who had BI-RADS-4 or BI-RADS-5 radiologic abnormalities (mean, 37.6 days vs 36.9 days; hazard ratio, 0.98; P ¼ .989). Timely diagnosis occurred more frequently among navigated Latinas (within 30 days: 67.3% vs 57.7%; P ¼ .045; within 60 days: 86.2% vs 78.4%; P ¼ .023). This was driven by the BI-RADS-3 strata (within 30 days: 83.6% vs 50%; P < .001; within 60 days: 94.5% vs 67.2%; P < .001). A lack of missed appointments was associated with timely diagnosis. CONCLUSIONS. Patient-centered navigation to assist Latina women with abnormal screening mammograms appeared to reduced the time to diagnosis and increase rates of timely diagnosis overall. However, in stratified analyses, only navigated Latinas with an initial BI-RADS-3 screen benefited, probably because of a reduction in missed diagnostic appointments in this group.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking female Hispanics over 18 years of age who attend this clinic and who receive mammography screening results specified as BI-RADS 3, 4 or 5, will be offered participation in the study.
* Although not actively recruited, pregnant women will not be excluded from the study sample

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
T0-T1; Days from Index Screening to Diagnosis | 30 days
  Number of days from date of index screening abnormality to definitive diagnosis and the proportion achieving timely diagnosis (within 30 days or 60 days of screening).
T1-T2; Days from Diagnosis to Treatment Initiation | 30 days
  Number of days from date of definitive diagnosis to initiation of treatment and the proportion achieving timely treatment (within 30 or 60 days of diagnosis)

SECONDARY OUTCOMES:
# Barriers | 365 days
  Relationship of # of reported barriers by navigated women and relationship of it to T0-T1 and T1-T2
Patient Satisfaction | 365 days
  Patient satisfaction with navigation provided as measured by Patient Satisfaction scale
Mental Health Status | 365 days
  Patient mental health status pre- and post-navigation

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G Ramirez, DrPH, Principal Investigator — The University of Texas Health Science Center at San Antonio